CLINICAL TRIAL: NCT04508777
Title: COVID SAFE: COVID-19 Screening Assessment for Exposure
Acronym: COVID SAFE
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 843565-OBS
Record Dates: First submitted 2020-08-10; First posted 2020-08-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Covid19
Keywords: COVID-19; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Saliva-based testing — Participants will take part in a voluntary COVID-19 screening program that includes bi-weekly saliva-based testing.

SUMMARY:
In order to safely and effectively reopen businesses and universities across the US, institutions will need to develop approaches to rapidly identify COVID-19 cases and manage their spread while balancing program effectiveness, feasibility, costs, and scalability.

This study will evaluate the implementation of a COVID-19 screening program that coordinates several existing systems at the University of Pennsylvania including saliva-based viral testing.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) pandemic has resulted in close to 10,000,000 reported cases worldwide, including more than 2,000,000 aggregated reported cases and 120,000 deaths in the United States. Initial efforts to address the COVID-19 pandemic were aimed at testing symptomatic individuals, implementing stay-in-place orders, and at increasing hospital capacity to meet surge demands. While nations continue to confront the current crisis, plans for the future must be put in place tools to enhance our ability to conduct effective screening, containment, and case management.

Widespread COVID-19 testing is needed to safely and effectively reopen schools and businesses across the US. However, currently approved testing options require reagents that are limited in supply, severely hindering scalability. Emerging evidence indicates that saliva testing with the option of at-home sample collection can accurately identify COVID-19 viral infection. Additional diagnostic testing options will continue to increase patient access. Moreover, this approach provides an option for the easy, safe and convenient collection of samples required for testing without traveling to a doctor's office, hospital, or testing site. Collection by the patient also reduces exposure of health care workers to the virus and preserves limited personal protective equipment.

With access to expanded testing, health systems and universities will need to test alternative methods to manage COVID-19 spread while balancing program effectiveness, feasibility, costs, and scalability. Insights from the field of behavioral economics offer promise for designing and sustaining these kinds of policies. For these reasons, the investigators propose to evaluate the implementation of a COVID-19 screening program that uses saliva-based testing.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* University of Pennsylvania faculty, staff, or trainee
* Have a phone or device capable of receiving text messages
* Willing to participate in the study for 6 months

Exclusion Criteria:

* Participants will not be eligible if they identify any reason they are unable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of University of Pennsylvania faculty, staff, and trainees
Sampling Method: Non-Probability Sample
Enrollment: 1759 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Test compliance | 3 months
  The rate of compliance with saliva-based testing

OTHER OUTCOMES:
Test compliance | 6 months
  The rate of compliance with saliva-based testing

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh S Patel, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States